CLINICAL TRIAL: NCT00243503
Title: A Phase 2 Efficacy And Safety Study Of SU011248 In Combination With Trastuzumab As Treatment For Metastatic Disease In Patients With Breast Cancer
Brief Title: Open Label Study Of SU011248 In Combination With Trastuzumab For Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181067
Record Dates: First submitted 2005-10-20; First posted 2005-10-24 (Estimated); Results first posted 2010-05-19 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer Metastatic
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: SU011248/Trastuzumab

INTERVENTIONS:
Drug: SU011248/Trastuzumab — SU011248 will be administered orally, starting dose of 37.5 mg daily on a continuous regimen. Trastuzumab will be administered weekly (loading dose 4 mg/kg followed by weekly 2mg/kg) or every 3 weeks (loading dose 8 mg/kg followed by 6mg/kg q3w). Study treatment should continue until progression, withdrawal for other reasons, or for up to 18 months following which patients requiring continued access will be offered SU011248 on a separate protocol.

SUMMARY:
The current study is to evaluate: Overall response rate for the combination of trastuzumab and SU011248 in metastatic or locally recurrent breast cancer; evaluate safety and tolerability of the combination; measure duration of tumor control and survival; assess patient reported outcomes; assess PK in combination with trastuzumab and compare efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of breast cancer with evidence of 1) unresectable, locally recurrent, or 2) metastatic disease.
* HER2 positive disease (3+ by immunohistochemistry [IHC] or FISH-positive)
* Candidate for treatment with trastuzumab. Prior treatment with trastuzumab and or/ lapatinib in the neoadjuvant, adjuvant or metastatic disease setting is permitted. Treatment with hormone therapy in the adjuvant and/or advanced disease setting is permitted.

Exclusion Criteria:

* Prior treatment with >1 regimen of cytotoxic therapy in the advanced disease setting. Adjuvant chemotherapy is permitted
* Prior exposure to trastuzumab if the patient had developed severe hypersensitivity reactions.
* Prior treatment on a SU11248 clinical trial.
* Uncontrolled brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (14):
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Harvey, Illinois
  - Pfizer Investigational Site, Tinley Park, Illinois
  - Pfizer Investigational Site, Munster, Indiana
  - Pfizer Investigational Site, Lafayette, Louisiana
  - Pfizer Investigational Site, New Iberia, Louisiana
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Memphis, Tennessee
- Belgium (2):
  - Pfizer Investigational Site, Ottignies
  - Pfizer Investigational Site, Wilrijk
- Canada (3):
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Greenfield Park, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- France (3):
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Saint-Cloud
- Spain (3):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Valencia, Valencia

REFERENCES:
- [Derived] Bachelot T, Garcia-Saenz JA, Verma S, Gutierrez M, Pivot X, Kozloff MF, Prady C, Huang X, Khosravan R, Wang Z, Cesari R, Tassell V, Kern KA, Blay JY, Lluch A. Sunitinib in combination with trastuzumab for the treatment of advanced breast cancer: activity and safety results from a phase II study. BMC Cancer. 2014 Mar 7;14:166. doi: 10.1186/1471-2407-14-166. PMID 24606768
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181067&StudyName=Open%20Label%20Study%20Of%20SU011248%20%20In%20Combination%20With%20Trastuzumab%20For%20Patients%20With%20Metastatic%20Breast%20Cancer%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab + Sunitinib: Trastuzumab was administered intravenously (i.v) weekly (loading 4 mg/kg followed by weekly 2 mg/kg) or every 3 weeks (loading 8 mg/kg followed by 6 mg/kg thrice weekly). Sunitinib began with 37.5 mg by oral capsule once daily in a continuous regimen. Treatment was administered in 4-week cycles.
Period: Overall Study
Arm/Group | Trastuzumab + Sunitinib
Started | 60 (3 participants discontinued and only took Trastuzumab.)
Completed | 2
Not Completed | 58
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 44
Not completed — Death | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 60
Age Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
EORTC QLQ-C30 [Mean (Standard Deviation); unit: scores on a scale] — European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30).Response range:not at all-very much,global/QOL range:very poor-excellent.Scale/single-item-score 0-100.Higher functional/global=better functioning and symptom=greater degree of symptoms.'n' = participants evaluated at timepoint for each group.
  scores on a scale
    Function Score: Global health (n=48) | 66.8 (26.8)
    Function Score: Physical function (n=49) | 79.5 (21.3)
    Function Score: Role function (n=49) | 76.2 (30.0)
    Function Score: Cognitive function (n=49) | 82.0 (25.6)
    Function Score: Emotional function (n=49) | 62.8 (26.4)
    Function Score: Social function (n=49) | 75.5 (29.9)
    Symptom Score: Fatigue (n=49) | 35.6 (27.6)
    Symptom Score: Pain (n=49) | 38.8 (33.7)
    Symptom Score: Nausea/vomiting (n=49) | 7.1 (18.0)
    Symptom Score: Dyspnea (n=48) | 22.9 (28.5)
    Symptom Score: Loss of appetite (n=49) | 14.3 (28.1)
    Symptom Score: Insomnia (n=49) | 35.4 (31.5)
    Symptom Score: Constipation (n=48) | 18.1 (32.9)
    Symptom Score: Diarrhea (n=49) | 6.8 (15.2)
    Symptom Score: Financial difficulty (n=48) | 15.3 (28.3)
EORTC QLQ Breast Cancer Module (BR23) [Mean (Standard Deviation); unit: scores on a scale] — EORTC QLQ (BR23): consist of 23 questions. Response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
  The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
  scores on a scale
    Function Score : Body image (n=46) | 77.2 (25.4)
    Function Score: Sexual function (n=44) | 21.6 (24.5)
    Function Score: Sexual enjoyment (n=15) | 53.3 (21.1)
    Symptom Score: Arm (n=48) | 23.8 (25.3)
    Symptom Score: Breast (n=47) | 25.9 (27.5)
    Symptom Score: systemic therapy side effects(n=48) | 17.2 (17.4)
    Others :Upset of hair loss (n=6) | 50.0 (27.9)
    Others :Future health perspective (n=48) | 39.6 (32.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Confirmed Objective Disease Response
Description: Objective disease response =participants with confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). A CR was defined as the disappearance of all target and non-target lesions. A PR was defined as a > = 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions associated to a non-progressive disease response for the non target lesions.
Time Frame: From start of treatment through 18 months
Population: The intent-to-treat (ITT) population included all enrolled participants who were treated with the combination (trastuzumab and sunitinib).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 57
percentage of participants | 36.8 [24.4 to 50.7]

2. Secondary Outcome: Duration of Response (DR)
Description: Time from the first documentation of objective tumor response (CR or PR) that was subsequently confirmed to the first documentation of objective tumor progression or death due to any cause. If tumor progression data included more than 1 date, the first date was used. DR was calculated as (the end date for DR minus first CR or PR that was subsequently confirmed +1) divided by 7.
Time Frame: From start of treatment through 18 months
Population: DR was calculated for the subgroup of participants from the ITT set, with a confirmed objective tumor response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 21
weeks | 25.6 [22.4 to 32.9]

3. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Percent of participants with confirmed CR, PR or stable disease (SD) for at least 24 weeks on study according to RECIST.CR was defined as disappearance of all target and non-target lesions.PR was defined as >=30% decrease in sum of longest dimensions of target lesions taking as reference baseline sum longest dimensions associated to non-progressive disease response for non target lesions.SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference smallest sum of longest dimensions since treatment started.
Time Frame: From start of treatment through 18 months
Population: The ITT population included all enrolled participants who were treated with the combination (trastuzumab and sunitinib).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 57
Percentage of Participants | 56.1 [42.4 to 69.3]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from first dose of study treatment to first documentation of objective tumor progression, or to death on-study due to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. PFS was calculated as (first event date minus first dose date +1) divided by 7.
Time Frame: From start of treatment through 18 months
Population: The ITT population included all enrolled participants who were treated with the combination (trastuzumab and sunitinib).
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 57
Weeks | 28.0 [24.1 to 31.3]

5. Secondary Outcome: Time to Progression (TTP)
Description: Time from first dose of study treatment to first documentation of objective tumor progression. If tumor progression data included more than 1 date, the first date was used. TTP was calculated as (first event date minus first dose date +1) divided by 7.
Time Frame: From start of treatment through 18 months
Population: The ITT population included all enrolled participants who were treated with the combination (trastuzumab and sunitinib).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 57
weeks | 26.0 [23.3 to 31.1]

6. Secondary Outcome: Overall Survival (OS)
Description: Time from first dose of study treatment to first documentation of death due to any cause. OS was calculated as (date of death minus first dose date +1) divided by 7 * 4.33.
Time Frame: From start of study treatment until death or 2 years from first study treatment
Population: The ITT population included all enrolled participants who were treated with the combination (trastuzumab and sunitinib).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 57
months | NA [NA to NA] — Median OS was not reached.

7. Secondary Outcome: Probability of Survival at One Year
Description: One- year survival probability was estimated using the Kaplan-Meier method.
Time Frame: From start of study treatment until death or 2 years from first study treatment
Population: The ITT population included all enrolled participants who were treated with the combination (trastuzumab and sunitinib).
Measure: Number (95% Confidence Interval); unit: percentage of 1-year survival
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 57
percentage of 1-year survival | 91.2 [80.2 to 96.3]

8. Secondary Outcome: EORTC QLQ-C30
Description: EORTC QLQ-C30 scales consist of 30 questions: functional (physical/role/cognitive/emotional/ social), symptom (fatigue/nausea/vomiting/pain), global health/QOL, cancer symptom (dyspnea/insomnia/appetite loss/constipation/diarrhea). Feelings in past week: response range: not at all to very much, global/QOL range: very poor to excellent. Scales/single-items averaged, score 0 to 100. Higher functional/global=better functioning and symptom=greater degree of symptoms.
Time Frame: From start of treatment through 18 months
Population: The ITT population included all enrolled participants who were treated with the combination (trastuzumab and sunitinib).The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 57
scores on a scale
  Function Score: Global health (n=28) | 56.0 (21.4)
  Function Score: Physical function (n=28) | 75.2 (16.8)
  Function Score: Role function (n=28) | 60.1 (28.8)
  Function Score: Cognitive function (n=28) | 84.5 (21.7)
  Function Score: Emotional function (n=28) | 66.1 (27.5)
  Function Score: Social function (n=28) | 66.7 (28.3)
  Symptom Score: Fatigue (n=28) | 45.0 (25.3)
  Symptom Score: Pain (n=28) | 36.9 (25.8)
  Symptom Score: Nausea/vomiting (n=28) | 6.5 (10.5)
  Symptom Score: Dyspnea (n=28) | 26.2 (30.6)
  Symptom Score: Loss of appetite (n=28) | 20.2 (24.6)
  Symptom Score: Insomnia (n=28) | 29.8 (27.7)
  Symptom Score: Constipation (n=27) | 14.8 (26.7)
  Symptom Score: Diarrhea (n=27) | 32.1 (32.7)
  Symptom Score: Financial difficulty (n=28) | 17.9 (29.4)

9. Secondary Outcome: EORTC QLQ (BR23)
Description: BR23: consisted of 23 questions which measured disease related symptoms of dry mouth, eye pain, hair loss, hot flushes, attractiveness, future health, sexual activity, arm/shoulder pain, breast pain, swollen breast, and skin problems on the breast. Recall period: past week; response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
Time Frame: From start of treatment through 18 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 57
scores on a scale
  Function Score : Body image (n=27) | 76.4 (29.5)
  Function Score: Sexual function (n=24) | 14.6 (16.5)
  Function Score: Sexual enjoyment (n=10) | 33.3 (15.7)
  Others :Future health perspective (n=27) | 45.7 (34.8)
  Symptom Score: systemic therapy side effects(n=27) | 21.7 (15.8)
  Symptom Score: Breast (n=27) | 19.4 (23.6)
  Symptom Score: Arm (n=27) | 21.0 (23.9)
  Others :Upset of hair loss (n=6) | 44.4 (27.2)

10. Secondary Outcome: Dose-corrected Trough Plasma Concentrations (Ctrough) of Sunitinib
Description: Ctrough = the concentration prior to study drug administration. Dose-corrected values were reported, the reference dose was 37.5 mg.
Time Frame: Predose on Day 1 of Cycle 3 and 5
Population: The Pharmacokinetic (PK) population included all enrolled participants who were treated with the combination (trastuzumab and sunitinib) and collected plasma values.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 47
nanograms (ng)/milliliter (mL)
  Day 1 (Cycle 3) | 53.5 (27.6)
  Day 1 (Cycle 5) | 55.0 (24.8)

11. Secondary Outcome: Dose-corrected Ctrough of SU-012662 (Sunitinib's Metabolite)
Description: as for outcome 10
Time Frame: Predose on Day 1 of Cycle 3 and 5
Population: The PK population included all enrolled participants who were treated with the combination (trastuzumab and sunitinib) and collected plasma values.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 47
ng/mL
  Day 1 (Cycle 3) | 26.7 (14.4)
  Day 1 (Cycle 5) | 24.7 (12.5)

12. Secondary Outcome: Dose-corrected Ctrough of Total Drug (Sunitinib + SU-012662)
Description: as for outcome 10
Time Frame: Predose on Day 1 of Cycle 3 and 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Trastuzumab + Sunitinib
Number analyzed (Participants) | 47
ng/mL
  Day 1 (Cycle 3) | 80.2 (39.9)
  Day 1 (Cycle 5) | 79.7 (36.3)

ADVERSE EVENTS:
Time Frame: From time of informed consent signing (SAEs) or first study treatment (AEs) through 18 months and including 28 calendar days after the last dose of study drug.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Trastuzumab + Sunitinib
Serious Adverse Events (participants affected / at risk) | 25/60
Other Adverse Events (participants affected / at risk) | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Sunitinib (N=60)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Periodontal disease (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Multi-organ failure (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Ejection fraction decreased (Investigations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
Drug interaction (General disorders) | 1
Device related infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Sunitinib (N=60)
Anaemia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Left ventricular dysfunction (Cardiac disorders) | 10
Hypothyroidism (Endocrine disorders) | 5
Eyelid oedema (Eye disorders) | 6
Lacrimation increased (Eye disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 36
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 20
Gingival bleeding (Gastrointestinal disorders) | 4
Gingival pain (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 20
Rectal haemorrhage (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 21
Asthenia (General disorders) | 29
Chest pain (General disorders) | 3
Chills (General disorders) | 5
Fatigue (General disorders) | 19
Mucosal inflammation (General disorders) | 21
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 4
Pyrexia (General disorders) | 11
Nasopharyngitis (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 3
Ejection fraction decreased (Investigations) | 13
Electrocardiogram QT prolonged (Investigations) | 3
Weight decreased (Investigations) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dysgeusia (Nervous system disorders) | 27
Headache (Nervous system disorders) | 18
Paraesthesia (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 9
Chromaturia (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 15
Erythema (Skin and subcutaneous tissue disorders) | 6
Hair colour changes (Skin and subcutaneous tissue disorders) | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 9
Skin discolouration (Skin and subcutaneous tissue disorders) | 3
Yellow skin (Skin and subcutaneous tissue disorders) | 13
Haematoma (Vascular disorders) | 3
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 25
Vertigo (Ear and labyrinth disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 3
Cheilitis (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 3
Blood alkaline phosphatase increased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.